CLINICAL TRIAL: NCT03330353
Title: Functional Assessment of the Melanopsin-Containing Retinal Ganglion Cells in Progressive Supranuclear Palsy Using Chromatic Pupillometry
Brief Title: Chromatic Pupillometry to Assess the Melanopsin-Light Pathway in Progressive Supranuclear Palsy
Acronym: PMPSP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: NeurOptics Inc. (Industry); University of Toronto (Other)
Responsible Party: Principal Investigator, Shirley Wray, Professor of Neurology, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2017p001603
Record Dates: First submitted 2017-09-19; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: PSP - Progressive Supranuclear Palsy; PD - Parkinson's Disease; AD - Alzheimer's Disease; ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Parkinson Disease; Alzheimer Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurodegenerative Diseases: Individuals with neurodegenerative diseases
  Interventions: Diagnostic Test: Pupillometry

INTERVENTIONS:
Diagnostic Test: Pupillometry — Use of pupillometry to assess melanopsin-light pathway in patients with neurodegenerative diseases

SUMMARY:
The specific aim of this study is to investigate rod, cone and melanopsin driven pupillary light response in individuals with progressive supranuclear palsy (PSP), age-matched healthy controls and individuals with other neurodegenerative diseases using chromatic pupillometry, with special interest in assessing melanopsin-driven post-illumination pupil response (PIPR) as an identifier for PSP.

The study addresses the following hypotheses:

1. Chromatic pupil responses, including rod/cone-driven rapid phase constriction and melanopsin-driven PIPR, are reduced in subjects with PSP compared to age-matched normal healthy control subjects,
2. Pupil parameters of the melanopsin-driven PIPR are abnormal in PSP subjects without supranuclear palsy, which is indicative of a subclinical physiological deficit of the OPN in the early stages of PSP.

If these hypotheses are upheld, chromatic pupillometry to measure the PIPR promises to be a reliable in vivo, non-invasive, convenient and inexpensive technique to detect asymptomatic pupillomotor impairment in advance of diagnostic oculomotor signs and deterioration of cognitive function.

DETAILED DESCRIPTION:
In 1963, Richardson, Steele and Olszewski published a landmark clinical report on 8 cases of supranuclear ophthalmoplegia, pseudobulbar palsy, nuchal dystonia and dementia and established the syndrome of heterogeneous system degeneration as a clinicopathological entity now known as PSP. The disease has a characteristic onset in the sixth decade (range 45 to 75 years) with some combination of impaired balance, abrupt falls, visual disturbances, slurred speech, dysphasia and vague changes in personality.

Slowing of voluntary vertical saccades, either down, up or both are a diagnostic marker of PSP and later impairment of voluntary horizontal saccades are characteristic in more than half of the cases. However, a proportion of PSP patients do not demonstrate these eye signs for a year or more after the onset of the disease.

This pilot study will use chromatic pupillometry to determine whether such a novel methodology may be used as an objective in vivo identifier of PSP. The rationale for the study is based in part on:

1. Clinicopathological correlation between the key clinical signs of a supranuclear gaze palsy with pathological verification that the degenerative process affects the pretectum and rostral midbrain,
2. The melanopsin-signaling pathway from ipRGCs (intrinsically photosensitive retinal ganglion cells) in the eye projects to the OPN (olivary pretectal nucleus) in the midbrain,
3. Chromatic pupillometry is a non-invasive technique suitable for elderly subjects with or without dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals that meet the clinical criteria for PSP. Core features include:

   * Recurrent falls and unsteady gait
   * Axial and nuchal rigidity
   * Pseudobulbar palsy
   * Bilateral lid retraction
   * Supranuclear vertical gaze palsy
   * Atrophy of the midbrain tegmentum (the hummingbird sign on brain MRI,
2. Individuals that fit the criteria for the second PSP phenotype (which resembles PD) that has asymmetric findings, tremors and poor responses to treatment with Levodopa,
3. Individuals that meet the clinical criteria for PD with:

   * Progressive bradykinesia
   * Postural instability and frequent falls
   * Festinating gait with loss of associated movements
   * Cogwheel rigidity and mask-like face
   * Rest tremor,
4. Individuals who carry a diagnosis of Alzheimer' disease who present with progressive impairment of memory and cognitive domains such as language and visuospatial perception.

Diagnoses will be confirmed by the review of health/medical records of patients recruited from the Frontotemporal Disorders Unit clinic. In the case of participants recruited from research studies, diagnoses will be confirmed by the review of the research diagnoses indicated on the individuals' research records.

Exclusion Criteria:

1. Individuals who are frail or in questionable health,
2. Individuals with cataracts or with posterior pole ocular pathology such as age-related macular degeneration and optic neuropathies, including open angle high intraocular pressure glaucoma,
3. Individuals with photophobia (i.e., painful light sensitivity) when exposed to bright light, including those with ophthalmological conditions such as keratitis (herpes simplex), uveitis or Achromatopsia,
4. Individuals with advanced dementia with inability to sit erect, hold the eyes open, incontinence,
5. Individuals with epilepsy,
6. Individuals diagnosed with major depression or other severe psychiatric disorders

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with PSP and age-matched control subjects
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Pupil Constriction | 2 years
  The smallest pupil size following light stimulation. This parameter primarily represents rapid phase extrinsic ipRGC activity driven by rods and cones through synaptic input.
Post-illumination pupil response (PIPR) | 2 years
  Measured pupil diameter over a period of 20 seconds, from 10 to 30 seconds after the offset of light stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley H Wray, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Coded data will be shared with co-investigators

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT03330353/Prot_SAP_001.pdf
  • Informed Consent Form (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT03330353/ICF_002.pdf